CLINICAL TRIAL: NCT05068479
Title: Evaluation of the Safety & Efficacy of the Laser Scleral Microporation Procedure to Restore Visual Function and Range of Accommodation
Brief Title: Safety & Efficacy of the Laser Scleral Microporation Procedure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated early to pursue Gen II laser advancements
Sponsor: ACE Vision Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAN-AVG-PRES-2020-01
Record Dates: First submitted 2021-09-28; First posted 2021-10-05 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-08

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural Emmetropic Presbyopes (Experimental): Patients that did not undergo any vision correcting surgery or implantation of an intraocular lens but suffering from presbyopia will receive bilateral Laser Scleral Microporation procedure.
  Interventions: Device: Bilateral Laser Scleral Microporation procedure
- Post Laser Vision Correction (LVC) Emmetropic Presbyopes (Experimental): Patients that underwent laser vision correction procedure (e.g. LASIK) in the past and suffering from presbyopia will receive bilateral Laser Scleral Microporation procedure.
  Interventions: Device: Bilateral Laser Scleral Microporation procedure

INTERVENTIONS:
Device: Bilateral Laser Scleral Microporation procedure — Partial depth scleral microporations with an Er:YAG laser in a predetermined pattern.

SUMMARY:
A new minimally invasive procedure for treating presbyopia is being evaluated to determine if there is improvement in near and intermediate vision after treatment

DETAILED DESCRIPTION:
This is a prospective, controlled, single-center clinical study to evaluate the safety and efficacy of the Laser Scleral Microporation Procedure.

Laser Scleral Microporation Procedure is a treatment to restore visual and accommodative function in presbyopic patients. The subjects are bilaterally treated with the Laser Scleral Microporation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to understand and sign an informed consent;
2. Willing and able to adhere to the instructions set forth in this protocol;
3. 48 years of age or greater, of either gender or any race;
4. Less than (<) 1.00D of astigmatism in each eye, measured by manifest refraction;
5. Manifest refraction spherical equivalent refraction (MRSE) of less than or equal to +/- 0.50D for distance vision; Note: Subjects who meet this criterion as a result of prior laser refractive surgery may qualify; however, the subject must have had the Laser Vision Correction (LVC) at least 12 months prior to the LSM procedure and be stable.
6. Uncorrected distance visual acuity (UDVA) is better than or equal to 20/40 (logMAR 0.30) in each eye, and a Corrected Distance Visual Acuity (CDVA) is better than or equal to 20/25 (logMAR 0.10) in each eye;
7. Demonstrate Stereopsis of 100 seconds of arc or better using a Randot stereoscopic fly test with near correction;
8. In good ocular health with the exception of presbyopia;
9. Presbyopia as demonstrated by:

   1. Currently wearing reading glasses and/or bifocals with an ADD of +1.50D or more at 40cm in each eye; and
   2. Reduced near visual acuity at 40cm when corrected for distance (DCNVA) of 20/50 (logMAR 0.40) or worse in each eye; and
   3. Minimum non-adjusted NAVQ score of 10;
10. Intraocular pressure (IOP) >11mmHg and < 30 mmHg in each eye without IOP lowering medication;
11. Less than or equal to (≤) 0.50D difference between the manifest refraction spherical equivalent and the cycloplegic refraction spherical equivalent;
12. If the subject has had Laser Vision Correction (LVC) within 1-2 years prior to the LSM procedure, stable distance refraction is present, defined as ≤ 0.50D variation of refraction in the 12 months prior to the LSM procedure. Manifest refraction spherical equivalent cannot vary more than 0.50D from current spectacles that are at least 12 months of age, or from a documented refraction at least 12 months prior to the preoperative baseline exam; if baseline data is available.
13. Completed a washout period of two weeks (14 days) prior to LSM procedure from prior treatment with:

With prior medical clearance: non steroidal anti-inflammatory drugs (NSAIDs), blood thinners, aspirin, and other substances which may increase bleeding; Anti-oxidants, which could affect blood thinning: Any antioxidant supplements (e.g., Vitamin E, Acai, Ocuvite, greater than 1000mg of Omega-3, etc); Antioxidant food supplements, such as shitake mushroom, mushroom extract and oral antioxidants

Exclusion Criteria:

1. Self-reported current pregnancy or breast-feeding, or plans to become pregnant during the entire study period;
2. History of ocular trauma or prior ocular surgery, or expected to require retinal laser treatment or other ocular surgical intervention;
3. Presence of ocular pathology other than cataract such as:

   Amblyopia or strabismus Corneal abnormalities or disease History of Dry Eye treatments/devices (example: hot compresses, punctal plugs, automated or manual thermal expression, intense pulse light, nasolacrimal stimulation, thermal lid treatments, or any dry eye medications such as Cyclosporine, liftegrast, or topical steroids) Pupil abnormalities (e.g., corectopia, Adie's) Capsule or zonular abnormalities Intraocular inflammation Retinal/macular disease or pathology Glaucoma (any type)
4. History of prior ocular surgery, including:

   Previous corneal surgery (e.g. penetrating keratoplasty, DSEAK/DSEK/DMEK/ lamellar keratoplasty), except for LASIK, SMILE, EpiLASIK/LASEK, or PRK; Previous anterior or posterior chamber surgery (e.g., vitrectomy, laser iridotomy); Previous retinal surgery (e.g. retinal break, repair related to ocular trauma or detachment, or pathology that is likely to require surgical intervention such as lattice degeneration
5. Known pathology that may affect visual acuity and/or are predicted to cause future acuity losses to a level of 20/30 (logMAR 0.18) or worse (e.g., macular degeneration);
6. Keratoconus or keratoconus suspect with CDVA of less than (<) 20/20 (logMAR > 0.00) at distance;
7. Near visual acuity at 40cm equivalent to their distance vision with distance correction (i.e., no evident effect of reduced accommodative range);
8. Use of systemic or ocular medications that may affect vision (the use of any miotic or cycloplegic agent is specifically contraindicated);
9. Acute or chronic disease or illness that could increase the operative risk or confound the study outcome(s) (e.g., diabetes mellitus, immunocompromised, connective tissue disease);
10. Uncontrolled systemic or ocular disease;
11. Any abnormality preventing reliable applanation tonometry in EITHER eye;
12. Undilatable pupil such that one cannot examine the periphery of the retina;
13. Functional eye preference, defined as phoria measuring over 15dp horizontally and/or over 2dp vertically, any strabismus, or suppression.
14. History of scleral ectasia, scleritis, or episcleritis; or thin sclera < 400 microns, as determined by taking the average of three measurements with ultrasound biomicroscopy (UBM) pachymetry or optical coherence tomography (OCT);
15. History of nuclear sclerosis LOCS III grade 2 or worse and/or other cataracts reducing CDVA or (where measured at select sites) OSI > 2.5;
16. Known allergies tp study medications including topical steroids, antibiotics and NSAIDs;
17. Per Principal Investigator (PI) discretion, as described below:

Note: This above list of exclusion criteria is not all inclusive. Investigators should use medical judgement to exclude patients that have diseases/conditions which may compromise study results and/or patients that are not ideal candidates. Patient affect and/or expectations may be included in the evaluation of candidacy.

Min Age: 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Binocular Uncorrected Near Visual Acuity (UNVA) @40cm | 12 months postoperative
  Binocular UNVA is measured with ETDRS charts placed in 40cm distance. This assessment is done binocularly under photopic light conditions.

SECONDARY OUTCOMES:
Monocular Uncorrected Distance Visual Acuity (UDVA) @4m | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Monocular UDVA is measured with ETDRS charts placed in 4m distance. This assessment is done monocularly under photopic light conditions.
Binocular Uncorrected Distance Visual Acuity (UDVA) @4m | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Binocular UNVA is measured with ETDRS charts placed in 4m distance. This assessment is done monocularly under photopic light conditions.
Monocular Uncorrected Intermediate Visual Acuity (UIVA) @60cm | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Monocular UIVA is measured with ETDRS charts placed in 60cm distance. This assessment is done monocularly under photopic light conditions.
Binocular Uncorrected Intermediate Visual Acuity (UIVA) @60cm | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Binocular UIVA is measured with ETDRS charts placed in 60cm distance. This assessment is done binocularly under photopic light conditions.
Monocular Uncorrected Near Visual Acuity (UNVA) @40cm | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Monocular UNVA is measured with ETDRS charts placed in 40cm distance. This assessment is done monocularly under photopic light conditions.
Binocular Uncorrected Near Visual Acuity (UNVA) @40cm | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Binocular UNVA is measured with ETDRS charts placed in 40cm distance. This assessment is done binocularly under photopic light conditions.
Manifest refraction | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  The manifested refraction is measured by means of a phoropter. The data contains values for sphere, cylinder and axis of cylinder. This data will also be used to calculate the manifested refractive spherical equivalent (MRSE)
Monocular Best Corrected Distance Visual Acuity (CDVA) @4m | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Monocular CDVA is measured with ETDRS charts placed in 4m distance using best aided corrective glasses. This assessment is done monocularly under photopic light conditions.
Binocular Best Corrected Distance Visual Acuity (CDVA) @4m | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Binocular CDVA is measured with ETDRS charts placed in 4m distance using best aided corrective glasses. This assessment is done binocularly under photopic light conditions.
Monocular Distance Corrected Intermediate Visual Acuity (DCIVA) @60cm | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Monocular DCIVA is measured with ETDRS charts placed in 60cm distance using corrective glasses for far distance. This assessment is done monocularly under photopic light conditions.
Binocular Distance Corrected Intermediate Visual Acuity (DCIVA) @60cm | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Binocular DCIVA is measured with ETDRS charts placed in 60cm distance using corrective glasses for far distance. This assessment is done binocularly under photopic light conditions.
Monocular Distance Corrected Near Visual Acuity (DCNVA) @40cm | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Monocular DCNVA is measured with ETDRS charts placed in 40cm distance using corrective glasses for far distance. This assessment is done monocularly under photopic light conditions.
Binocular Distance Corrected Intermediate Near Acuity (DCNVA) @40cm | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Binocular DCNVA is measured with ETDRS charts placed in 40cm distance using corrective glasses for far distance. This assessment is done binocularly under photopic light conditions.
Determination of reading prescription | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Reading prescription is determined by using refraction for fars distance, placing ETDRS charts in 40cm distance and adding positive lenses to the refraction glasses until further addition of positive lenses has no more effect on the reading ability of the subject. The added positive lenses (in diopter) is noted down in the CRF.
Monocular Best Corrected Near Visual Acuity (CNVA) @40cm | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Monocular CNVA is measured with ETDRS charts placed in 40cm distance using corrective glasses for near distance (reading prescription). This assessment is done monocularly under photopic light conditions.
Accommodative Amplitude using binocular minus lens to blur | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  The amplitude of accommodation will be assessed binocularly at distance with an introduction of minus power over the distance prescription to stimulate accommodation. Instruct the patient to focus on the distance vision chart, and slowly add minus power in -0.25D steps until the subject reports first sustained blur on the line. Record the dioptric value where the subject reports the first sustained blur. Subtract the distance prescription from this value to obtain the accommodative amplitude using this method. This test is repeated three times. This assessment is done monocularly under photopic light conditions.
Accommodative Amplitude using monocular minus lens to blur | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  The amplitude of accommodation will be assessed monocularly at distance with introduction of minus power over the distance prescription to stimulate accommodation. Place an occluder lens into the trial frame over the left eye. Instruct the patient to focus on the distance vision chart and slowly add minus power in -0.25D steps until the subject reports first sustained blur on the line. Record the dioptric value where the subject reports the first sustained blur. Subtract the distance prescription from this value to obtain the accommodative amplitude using this method. This test is repeated three times. This assessment is done monocularly under photopic light conditions.
iReST reading test | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  The reading speed will be measured using the International Reading Speed Texts (iReST™), a standardized assessment of reading speed. For this test, the reading prescription determined at each visit will be used and the assessment will be done under photopic light conditions.
Accommodation testing | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  The iTrace (Tracey Technologies, Houston, TX or equivalent) wavefront aberrometer is used for the accommodation testing. The iTrace measures aberrometry at distance using the distance prescription in a trial frame, as well as at 60cm and 40cm using a near rod.
  Objective measures will be performed to assess the change in accommodation based upon the location of the visual target.
Wavefront measurement | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  The iTrace (Tracey Technologies, Houston, TX or equivalent) measures aberrometry at distance, 60cm and 40cm. Measurements will be performed unaided and aided using the distance prescription based upon the manifest refraction. Coma, Spherical Aberration, and Trefoil exams will also be recorded at distance, 60cm and 40cm.
Auto-Keratometry | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Simulated-keratometry (SimK) will be measured using the iTrace unit (Tracey Technologies, Houston, TX).
Corneal topography | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Anterior surface corneal topography using placido disc will be measured using the iTrace unit (Tracey Technologies, Houston, TX).
Corneal tomography | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 24 months postoperative
  Corneal tomography using Scheimpflug imaging will be measured using the Pentacam HR (Oculus, Wetzlar, Germany).
Stereoacuity | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Stereoacuity will be measured under photopic conditions using a standard randot stereoscopic test at 40cm with the subject's reading prescription.
  For this test, the reading prescription determined at each visit will be used and the assessment will be done under photopic light conditions.
Pupillometry under mesopic lighting conditions | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Measurement of pupil size will be performed under mesopic lighting conditions. The Neuroptics VIP® -200 pupillometer is being used for this assessment
Pupillometry under photopic lighting conditions | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Measurement of pupil size will be performed under photopic lighting conditions. The Neuroptics VIP® -200 pupillometer is being used for this assessment
Monocular contrast acuity | 1 month postoperative; 12 months postoperative; 24 months postoperative
  Contrast acuity will be measured using ETDRS optotypes with 10% contrast placed in 4m distance. For this test, best distance aided corrective glasses are used and this assessment is done monocularly under photopic light conditions.
Binocular contrast acuity | 1 month postoperative; 12 months postoperative; 24 months postoperative
  Contrast acuity will be measured using ETDRS optotypes with 10% contrast placed in 4m distance. For this test, best distance aided corrective glasses are used and this assessment is done binocularly under photopic light conditions.
Axial length measurement | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 24 months postoperative
  The axial length of the eye will be measured using a partial coherence interferometry device (IOLMaster version 7.5, Carl Zeiss Meditec).
Intraocular pressure measurement | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Intraocular Pressure will be measured using Goldmann applanation tonometry. Three measurements will be performed per eye at each visit.
Cycloplegic refraction | 12 months postoperative; 24 months postoperative
  A cycloplegic refraction at distance using 1% tropicamide will be performed. Following values will be recorded: sphere, cylinder, axis of cylinder.
Ultrasound biomicroscopy | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 24 months postoperative
  Ultrasonic Biomicroscopy (UBM) or OCT will be performed to assess scleral thickness and anatomical changes with accommodation. Three nonimmersion thickness measurements will be taken 4mm from the limbus (in any quadrant) to ensure the tissue thickness is sufficient for success and safety of the procedure.
Slitlamp examination | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of the eye structures.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  Corneal clarity anterior chamber cells anterior chamber flare lens grading using the LOCS III card Conjunctival/scleral vessel injection Degree of choroidal hue Conjunctival edema Conjunctival hemorrhages Eyelid edema
Dilated fundus exam | 12 months postoperative; 24 months postoperative
  A Dilated Fundus Exam will also be performed to examine the vitreous, optic nerve, blood vessels, macula and retina to identify eye related diseases or anatomical anomalies.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Jackson, MD, Study Director — Ace Vision Group
Locations (1):
- Panama Eye Center, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No